CLINICAL TRIAL: NCT00785941
Title: Phase I Study of Anti-Insulin-Like Growth Factor-I Receptor (IGF-IR) Monoclonal Antibody IMC-A12 Administered Every Other Week in Patients With Advanced Solid Tumors Who No Longer Respond to Standard Therapy or for Whom No Standard Therapy is Available
Brief Title: A Study of IMC-A12 Every 2 Weeks in Patients With Tumors Who No Longer Respond to Treatment or No Treatment is Available
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13933; CP13-0502 (Other: ImClone, LLC); I5A-IE-JAEI (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Advanced Solid Tumors
Keywords: Tumors; Antibodies, Monoclonal
MeSH Terms: conditions — Neoplasms | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-A12 (Experimental): All patients will receive intravenous infusions of IMC-A12, with the dose depending on which cohort they are enrolled into a minimum of three patients will be enrolled in each Cohort. When all patients complete a cohort, dose escalation to the next Cohort will occur.
  A treatment cycle will consist of IMC-A12 administered intravenously, once every other week for 4 weeks, for a total of 2 doses; followed by a 2-week observation period.
  Interventions: Biological: IMC-A12

INTERVENTIONS:
Biological: IMC-A12 — Cohort 1
  6 mg/kg I.V., once every other week for 4 weeks
  Other Names: Cixutumumab
Biological: IMC-A12 — Cohort 2
  10 mg/kg I.V., once every other week for 4 weeks
  Other Names: Cixutumumab
Biological: IMC-A12 — Cohort 3
  15 mg/kg I.V., once every other week for 4 weeks
  Other Names: Cixutumumab
Biological: IMC-A12 — Cohort 4
  21 mg/kg I.V., once every other week for 4 weeks
  Other Names: Cixutumumab
Biological: IMC-A12 — Cohort 5
  27 mg/kg I.V., once every other week for 4 weeks
  Other Names: Cixutumumab

SUMMARY:
The purpose of this study is to determine if IMC-A12 is safe for patients, and also to determine the best dose of IMC-A12 to give to patients.

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety profile and maximum tolerated dose (MTD) of the anti-IGF-IR monoclonal antibody IMC-A12 administered every other week in patients with advanced solid tumors who no longer respond to standard therapy or for whom no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria

* Patients with histopathologically-documented, measurable, advanced primary or recurrent solid tumors who no longer respond to standard therapy or for whom no standard therapy is available
* A life expectancy of >3 months
* Adequate hematologic function
* Adequate hepatic function
* Adequate renal function
* Use of effective contraception, if procreative potential exists.
* At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, prior radiation therapy (palliative radiation therapy is allowed), an open biopsy, or a significant traumatic injury to allow for adequate recovery
* At least 6 weeks must have elapsed from nitrosoureas, mitomycin C, or monoclonal antibody therapy to allow for adequate recovery
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center

Exclusion Criteria

* Any concurrent malignancy other than non-melanomatous skin cancer or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for ≥3 years will be allowed to enter the trial
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection requiring parenteral antibiotics
  * symptomatic congestive heart failure (class III or IV of the New York Heart Association classification for heart disease)
  * unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * uncontrolled hypertension (systolic blood pressure >160 mm Hg, diastolic blood pressure >100 mm Hg, found on two consecutive measurements separated by a 1-week period despite adequate medical support)
  * clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [National Cancer Institute {NCI}-Common Terminology Criteria for Adverse Events {CTCAE}, Version 3.0, grade 3] or asymptomatic sustained ventricular tachycardia)
  * psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements
  * patients with symptomatic brain metastases (patients with a history of brain metastases must be clinically stable and not taking steroids; anticonvulsants are allowed)
* A serious or nonhealing active wound, ulcer, or bone fracture
* Known human immunodeficiency virus-positive
* A history of a hemorrhagic or thrombotic disorder within 9 months
* Pregnant or breast feeding
* A history of prior treatment with other agents specifically targeting IGFRs.
* Known diabetes
* Inability or unwillingness to interrupt steroidal or hormonal therapy for the duration of treatment with IMC-A12
* A positive anti-IMC-A12 antibody response
* A history of allergic reactions to monoclonal antibodies or other therapeutic proteins
* Employees of the investigator or study center with direct involvement in this study or other studies under the direction of the investigator or study center, as well as family members of the employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 8 weeks
Maximum Tolerated Dose | 8 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax), cohorts 1, 2, 3, 4, and 5 | 8 weeks
Minimum concentration (Cmin), cohorts 1, 2, 3, 4, and 5 | 8 weeks
Area under concentration (AUC), cohorts 1, 2, 3, 4, and 5 | 8 weeks
Half-life (t 1/2), cohorts 1, 2, 3, 4, and 5 | 8 weeks
Clearance (Cl) rate drug is completely removed, cohorts 1, 2, 3, 4, and 5 | 8 weeks
Volume of distribution (Vss) at steady state, cohorts 1, 2, 3, 4, and 5 | 8 weeks
Serum Anti-IMC-A12 Antibody Assessment (immunogenicity) | 8 weeks
Change in tumor size from Baseline Measurement | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (1):
- ImClone Investigational Site, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Higano CS, Berlin J, Gordon M, LoRusso P, Tang S, Dontabhaktuni A, Schwartz JD, Cosaert J, Mehnert JM. Safety, tolerability, and pharmacokinetics of single and multiple doses of intravenous cixutumumab (IMC-A12), an inhibitor of the insulin-like growth factor-I receptor, administered weekly or every 2 weeks in patients with advanced solid tumors. Invest New Drugs. 2015 Apr;33(2):450-62. doi: 10.1007/s10637-015-0217-7. Epub 2015 Mar 7. PMID 25749986